CLINICAL TRIAL: NCT01535677
Title: A Bioequivalence Study of the Fixed Dose Combination Dapagliflozin/Metformin Tablet (5 mg/850 mg) Relative to a 5 mg Dapagliflozin Tablet and an 850 mg Metformin (Glucophage® Marketed in Canada by Sanofi-Aventis) Tablet Co-Administered to Healthy Subjects in the Fasted and Fed States
Brief Title: To Compare the Similarity of a Combination Dapagliflozin/Metformin Tablet With the Two Drugs Administered Separately
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D1691C00007
Record Dates: First submitted 2012-01-13; First posted 2012-02-20 (Estimated); Last update posted 2015-07-09 (Estimated); Status verified 2015-07

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Phase 1; healthy volunteers; cross-over study; Bioavailability; Bioequivalence; Cmax; tmax; AUC; AUC(0-t); λz; tlast
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin

ARMS (4):
- 1 (Experimental): 5 mg dapagliflozin and 850 mg Glucophage in fasted state
  Interventions: Drug: Dapagliflozin + Glucophage tablet fasted
- 2 (Experimental): dapagliflozin/metformin (5 mg/850 mg) immediate release (IR) FDC in fasted
  Interventions: Drug: Dapagliflozin/metformin IR FDC tablet fasted
- 3 (Experimental): 5 mg dapagliflozin and 850 mg Glucophage in fed state
  Interventions: Drug: Dapagliflozin + Glucophage tablet fed
- 4 (Experimental): dapagliflozin/metformin (5 mg/850 mg) IR FDC in fed state
  Interventions: Drug: Dapagliflozin/metformin IR FDC tablet fed

INTERVENTIONS:
Drug: Dapagliflozin + Glucophage tablet fasted — Single oral doses of 5 mg dapagliflozin and 850 mg Glucophage® tablets administered together in the fasted state
  Arms: 1
Drug: Dapagliflozin/metformin IR FDC tablet fasted — single oral dose of dapagliflozin/metformin (5 mg/850 mg) IR FDC tablet in the fasted state
  Arms: 2
Drug: Dapagliflozin + Glucophage tablet fed — Single oral doses of 5 mg dapagliflozin and 850 mg Glucophage® tablets administered together in the fed state
  Arms: 3
Drug: Dapagliflozin/metformin IR FDC tablet fed — single oral dose of dapagliflozin/metformin (5 mg/850 mg) IR FDC tablet in the fed state
  Arms: 4

SUMMARY:
This is an open-label, randomised study to compare the similarity of a combination Dapagliflozin/Metformin tablet with the two drugs administered separately under fasting and fed conditions in healthy volunteers.

DETAILED DESCRIPTION:
A Bioequivalence Study of the Fixed Dose Combination Dapagliflozin/Metformin Tablet (5.0 mg/850 mg) Relative to a 5.0 mg Dapagliflozin Tablet and an 850 mg Metformin (Glucophage® Marketed in Canada by Sanofi-Aventis) Tablet Co-Administered to Healthy Subjects in the Fasted and Fed States

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers aged 18 to 55 years inclusive with suitable veins for cannulation or repeated vein puncture
* Male subjects should be willing to use barrier contraception ie, condoms and spermicide, from the day of dosing until at least 3 months after dosing with the investigational product
* Non-pregnant, non-lactating female subjects who if pre-menopausal are using adequate birth control eg, oral, injectable, transdermal or implanted hormonal contraceptives, vaginal contraceptive ring, intrauterine device (IUD)/intrauterine systems
* Have a body mass index (BMI) between 18.5 and 30.0 kg/m2 inclusive (ie, within 15% of normal range) and weigh at least 50 kg and no more than 100 kg.

Exclusion Criteria:

* History or presence of gastrointestinal, hepatic or renal disease or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs
* Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG that may interfere with individual safety evaluation Current smokers who smoke more than 5 cigarettes per day (or equivalent use of tobacco products) or cannot give up smoking during the study
* Excessive intake of caffeine containing drinks eg, coffee, tea, caffeine containing energy drinks and cola (more than 5 cups of coffee or equivalent per day)
* Plasma donation within one month of screening or any blood donation/blood loss >500 mL during the 3 months prior to screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2013-04; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Area under the curve over the time (AUC) | pre-dose, 0.25 min, 0.5 min, 1h, 1.5h, 2 h, 3h , 4 h, 5 h , 6 h, 8 h, 10 h, 12 h, 16 h, 24 h, 30 h, 36 h, 42 h, 48 h, 54 h, 60 h and 72 h post-dose
  No statistical analysis will be performed
AUC from time zero to the time of last quantifiable analyte concentration (AUC(0-t)) | pre-dose, 0.25 min, 0.5 min, 1h, 1.5h, 2 h, 3h , 4 h, 5 h , 6 h, 8 h, 10 h, 12 h, 16 h, 24 h, 30 h, 36 h, 42 h, 48 h, 54 h, 60 h and 72 h post-dose
  No statistical analysis will be performed
Maximum concentration (Cmax) | pre-dose, 0.25 min, 0.5 min, 1h, 1.5h, 2 h, 3h , 4 h, 5 h , 6 h, 8 h, 10 h, 12 h, 16 h, 24 h, 30 h, 36 h, 42 h, 48 h, 54 h, 60 h and 72 h post-dose
  No statistical analysis will be performed

SECONDARY OUTCOMES:
Time to reach maximum analyte concentration (tmax) | pre-dose, 0.25 min, 0.5 min, 1h, 1.5h, 2 h, 3h , 4 h, 5 h , 6 h, 8 h, 10 h, 12 h, 16 h, 24 h, 30 h, 36 h, 42 h, 48 h, 54 h, 60 h and 72 h post-dose
  No statistical analysis will be performed
Terminal rate constant (λz) | pre-dose, 0.25 min, 0.5 min, 1h, 1.5h, 2 h, 3h , 4 h, 5 h , 6 h, 8 h, 10 h, 12 h, 16 h, 24 h, 30 h, 36 h, 42 h, 48 h, 54 h, 60 h and 72 h post-dose
  No statistical analysis will be performed
Time of last quantifiable analyte concentration (tlast) | pre-dose, 0.25 min, 0.5 min, 1h, 1.5h, 2 h, 3h , 4 h, 5 h , 6 h, 8 h, 10 h, 12 h, 16 h, 24 h, 30 h, 36 h, 42 h, 48 h, 54 h, 60 h and 72 h post-dose
  No statistical analysis will be performed
Terminal half-life (t1/2) | pre-dose, 0.25 min, 0.5 min, 1h, 1.5h, 2 h, 3h , 4 h, 5 h , 6 h, 8 h, 10 h, 12 h, 16 h, 24 h, 30 h, 36 h, 42 h, 48 h, 54 h, 60 h and 72 h post-dose
  No statistical analysis will be performed
Observed maximum analyte concentration (Cmax) | pre-dose, 0.25 min, 0.5 min, 1h, 1.5h, 2 h, 3h , 4 h, 5 h , 6 h, 8 h, 10 h, 12 h, 16 h, 24 h, 30 h, 36 h, 42 h, 48 h, 54 h, 60 h and 72 h post-dose
  No statistical analysis will be performed
Area under the plasma concentration-time curve from time zero extrapolated to infinity (AUC) | pre-dose, 0.25 min, 0.5 min, 1h, 1.5h, 2 h, 3h , 4 h, 5 h , 6 h, 8 h, 10 h, 12 h, 16 h, 24 h, 30 h, 36 h, 42 h, 48 h, 54 h, 60 h and 72 h post-dose
  No statistical analysis will be performed
Area under the plasma concentration-curve from time zero to the time of last quantifiable analyte concentration (AUC(0 t)) | pre-dose, 0.25 min, 0.5 min, 1h, 1.5h, 2 h, 3h , 4 h, 5 h , 6 h, 8 h, 10 h, 12 h, 16 h, 24 h, 30 h, 36 h, 42 h, 48 h, 54 h, 60 h and 72 h post-dose
  No statistical analysis will be performed
Elimination terminal half-life (t1/2) | pre-dose, 0.25 min, 0.5 min, 1h, 1.5h, 2 h, 3h , 4 h, 5 h , 6 h, 8 h, 10 h, 12 h, 16 h, 24 h, 30 h, 36 h, 42 h, 48 h, 54 h, 60 h and 72 h post-dose
  No statistical analysis will be performed
Safety profile description in term of Adverse Events | from first dose in treatment period 1 up to 10 days after final dose
  No statistical analysis will be performed
Safety profile description in term of Blood Pressure | at screening, once daily during the residential period (5 days each) and up to 10 days after final dose
  No statistical analysis will be performed
Safety profile description in term of Physical Examination | at screening, Day -1 and Day 4 at Visits 2 to 5 and up to 10 days after final dose
  No statistical analysis will be performed
Safety profile description in term of Electrocardiogram ECG | at screening and up to 10 days after final dose
  No statistical analysis will be performed
Safety profile description in term of Heart Rate | at screening, once daily during the residential period (5 days each) and up to 10 days after final dose
  No statistical analysis will be performed
Safety profile description in term of Safety Labs | at screening, on Day -1 and Day 4 (72 hours post-dose) at Visits 2 to 5 and up to 10 days after final dose
  No statistical analysis will be performed

CONTACTS AND LOCATIONS:
Overall Officials: Eva Johnsson, MD, Study Director — AstraZeneca Research and Development SE-431 83 Mölndal Sweden; Saeed Kahn, MBBS, Principal Investigator — Quintiles Drug Research Unit at Guy's Hospital, 6 Newcomen St, London SE1 1YR; Mirjana Kujacic, PHD, Study Chair — AstraZeneca Research and DevelopmentSE-431 83 Mölndal Sweden
Locations (1):
- Research Site, London, United Kingdom

REFERENCES:
- [Result] Chang M, Liu X, Cui D, Liang D, LaCreta F, Griffen SC, Lubin S, Quamina-Edghill D, Boulton DW. Bioequivalence, Food Effect, and Steady-State Assessment of Dapagliflozin/Metformin Extended-release Fixed-dose Combination Tablets Relative to Single-component Dapagliflozin and Metformin Extended-release Tablets in Healthy Subjects. Clin Ther. 2015 Jul 1;37(7):1517-28. doi: 10.1016/j.clinthera.2015.05.004. Epub 2015 Jun 3. PMID 26048185
- See also: D1691C00007_CSR_Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1195&filename=D1691C00007_CSR_Synopsis.pdf
- See also: D1691C00007_Clinical_Study_Protocol — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1195&filename=D1691C00007_Clinical_Study_Protocol_Redacted.pdf